CLINICAL TRIAL: NCT01540149
Title: Tel Aviv Sourasky MC Home Monitoring Registry
Brief Title: Tel Aviv Sourasky MC Home Monitoring Clinic Registry
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HMR_TelAviv_sourasky
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Home Monitoring With ICD Patient

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ICD implant

SUMMARY:
The purpose of the registry is to assess workload of a Home Monitoring based follow up for Biotronik implantable cardioverter defibrillators (ICD) and cardiac resynchronization therapy defibrillators (CRTD) patients.

DETAILED DESCRIPTION:
EP unit device clinic is a very busy clinic. Every 6 month the patients arrive for device follow up where the device parameters, patient condition and arrhythmic events are being reviewed, and reprogramming of the device (if needed) is done. Average net time of patient's stay in the clinic is between 30-45 minutes.

Patients implanted with the Lumax device family allows for a better automated follow up procedure via remote management (Home Monitoring).

ELIGIBILITY:
Inclusion Criteria:

* Approved indication for ICD or CRTD.
* Implanted with or replaced with a Biotronik Lumax device.
* Patient is willing and able to sign consent form.
* Willing and able to attend clinic visits and follow up schedule.
* Transmission of more than 80% at 3-month FU.
* Patient older than 18 years.

Exclusion Criteria:

* No indication for ICD or CRTD implant.
* Life expectancy shorter than 12 months.
* Pregnancy.
* Participation in other clinical studies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICD or CRTD implanted patient
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aharon Glik, MD, Principal Investigator — Tel Aviv Sourasky MC
Locations (1):
- Electrophisiology Department, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No